CLINICAL TRIAL: NCT07107282
Title: Evaluation of a Software to Predict the Postoperative Component Position in Total Hip Arthroplasty (THA): Accuracy of Predictions and Impact on Interoperative Placement in a Single Centre
Brief Title: Evaluation of a Software to Predict the Postoperative Component Position in Total Hip Arthroplasty (THA)
Status: Not yet recruiting | Type: Observational
Sponsor: Marcel Jakob (Other)
Collaborators: Basel Academy for Quality and Research in Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Marcel Jakob, Prof. Dr., crossklinik AG
Organization: crossklinik AG (Other)
Other Study IDs: VerifierVerifier
Record Dates: First submitted 2025-07-16; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Total Hip Arthroplasty
Keywords: implant position; leg length

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All patients: All patients included in the study
  Interventions: Device: MyHip Verifier

INTERVENTIONS:
Device: MyHip Verifier — Numerical information on the position of the implant is provided to the surgeon.

SUMMARY:
The goal of this observational study is to learn about the accuracy of a software determining the implant position during THA surgery.

Measurements made with the software are compared to reference values determined on X-rays.

DETAILED DESCRIPTION:
The software is based on comparing an pre-operative fluoroscopy-based image with inter-operative fluoroscopy-based image. Three numerical values are provided: "leg length", "lateral offset" and "inclination".

Correponding reference values are determined based on pre-operative and post-operative X-rays.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for THA
2. Age of 18 or above

Exclusion Criteria:

1. Patients with anatomical conditions which reduce the applicability of the software
2. Patients with implants which reduce the applicability of the software
3. Patients who cannot perform an upright X-ray

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total hip arthrosplasty
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mean absolute difference between measured value and reference value | This measure involves two time points: Stopping of the software during surgery and performing the postoperative X-ray. The latter is usually the first day after surgery. A delay is allowed if a patient cannot perform an upright X-ray.
  The mean absolute difference between the final value measured by the software and the reference value determined on a postoperative X-ray.

SECONDARY OUTCOMES:
Mean amount of repositioning performed by the surgeon | This measure involves two time points: Starting and stopping of the software during surgery.
  The mean absolute difference between the value measured by the software when started and the final value
Mean absolute improvement in reaching the target value | This measure involves three time points: Determining target values prior to surgery and starting and stopping the software during surgery,
  The mean value of the change in absolute difference between the actual position and the target value from starting the software until stopping the software.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Jakob, MD, Principal Investigator — crossklinik AG

IPD SHARING:
Plan to Share IPD: Yes
An anonymized version of the statistical analysis data set will be published as part of the main publication.
Supporting Information: Study Protocol
Time Frame: IPD will be available at the date of publication of the main manuscript.
Access Criteria: There are no access criteria.